CLINICAL TRIAL: NCT06570408
Title: Precision Application of Clostridium Butyricm of Clinical Research on Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC3-047
Record Dates: First submitted 2024-07-29; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis; Knee
Keywords: Clostridium butyricum; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (placebo) (Placebo Comparator)
  Interventions: Behavioral: Western Ontario and McMaster University Osteoarthritis Index (WOMAC); Behavioral: Visual Analogue Scale (VAS); Diagnostic Test: Kellgren Lawrence Grading Scale (KL score); Behavioral: Quality of Life Questionnaires and Assessments:
- Group B (Treatment) (Experimental)
  Interventions: Behavioral: Western Ontario and McMaster University Osteoarthritis Index (WOMAC); Behavioral: Visual Analogue Scale (VAS); Diagnostic Test: Kellgren Lawrence Grading Scale (KL score); Behavioral: Quality of Life Questionnaires and Assessments:

INTERVENTIONS:
Behavioral: Western Ontario and McMaster University Osteoarthritis Index (WOMAC) — 1. WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales
Behavioral: Visual Analogue Scale (VAS) — 2. VAS is one of the pain rating scales used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Diagnostic Test: Kellgren Lawrence Grading Scale (KL score) — 3. KL score is the most widely used clinical tool for the radiographic diagnosis of OA.Each radiograph was assigned a grade from 0 to 4,
Behavioral: Quality of Life Questionnaires and Assessments: — 4. Quality of Life Questionnaires and Assessments: include quality of life, intestinal tract, conscious assessment of pain relief.etc.

SUMMARY:
Osteoarthritis (OA) is a common joint disease worldwide. The main symptom is that the mechanical wear of the cartilage in the joint and leads to the abnormal proliferation of the surrounding bone and synovial tissue with the chronic inflammation and the narrowing of the joint cavity. The prevalence of OA is increasing due to population increasing and aging, and there are currently about 400 million OA patients in worldwide. The treatment methods of osteoarthritis are mainly divided into medicine and non-medicine therapy. The major function of medicine therapy is to reduce pain and the arthroscopic surgery (arthroscopy) is main treatment of non-medicine therapy. Thus, in this project the investigators will mainly focus on the precise application of Clostridium butyricum on OA and the investigators' previous study successfully demonstrated the therapeutic effects of Clostridium butyricum on OA animal model. Therefore, will test the clinical effects of OA patient with Clostridium butyricum treatment, and whether it is also possible to improve the symptom of OA patients.

ELIGIBILITY:
Inclusion Criteria:

- A. Patients aged 55 to 75 years old with degenerative arthritis, diagnosed by a physician as suitable for participation in this experiment.

B. Patients with early-stage degenerative arthritis symptoms, as interpreted by X-ray using the Kellgren Lawrence Grading Scale at grade 1 or 2, and determined by a physician to not require long-term treatment.

C. Patients with a high pain index when the knee is extended 40-70 mm.

D. Patients who feel knee pain, primarily those with a high Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index score (pain scale score >2.0 or total WOMAC scale score >12).

Exclusion Criteria:

- A. Patients with a history of knee joint trauma or knee joint surgery (including arthroscopic surgery).

B. Patients who have taken steroid medication for the treatment of degenerative arthritis.

C. Patients with severe cardiovascular, cerebrovascular, rheumatic, or psychiatric diseases.

D. Patients with joint pain caused by other factors.

E. Patients with infectious diseases or acute infections (e.g., fever, localized inflammation, abscess).

F. Patients with systemic or metabolic diseases, or progressive bone degeneration caused by medication.

G. Cancer patients.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Day 0, 7, 14, 30, 60, 90
  used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales. The maxima score is 105, which have more high score mean more severe level of osteoarthritis.
Visual Analogue Scale (VAS) | Day 0, 7, 14, 30, 60, 90
  one of the pain rating scales used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. The minima score is 0. The maxima score is 10 for each knee. the higher score mean patient feel more pain on knee joint.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided